CLINICAL TRIAL: NCT05324462
Title: Glycaemic Control and Other Clinical Parameters in Adult Type 2 Diabetes Patients on Basal Insulin Initiating Treatment With IDegLira in Routine Clinical Practice in Colombia - A Single-arm, Non-interventional Retrospective Chart Review Study
Brief Title: Glycaemic Control and Other Clinical Parameters in Adult Type 2 Diabetes Patients on Basal Insulin Initiating Treatment With IDegLira in Routine Clinical Practice in Colombia
Acronym: SPIRIT
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9068-4884; U1111-1266-5484 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-04-04; First posted 2022-04-12 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — IDegLira

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IDegLira: Adult patients with T2D who have initiated treatment with IDegLira a minimum of 26 weeks
  Interventions: Drug: IDegLira

INTERVENTIONS:
Drug: IDegLira — Collecting data reported in medical records of patients with T2D, who had initiated treatment with commercially available IDegLira according to the routine clinical practice and local label at the discretion of the treating physician

SUMMARY:
The purpose of this study is to investigate the glycaemic control and other clinical parameters in adult patients previously treated with basal insulin (with or without OADs) and switched to IDegLira in real-world clinical practice in Colombia.

ELIGIBILITY:
Inclusion criteria:

1. Male or female, age above or equal to 18 years at the time of data collection.
2. Patient diagnosed with T2D greater than or equal to 12 months prior to data collection.
3. The decision to initiate treatment with commercially available IDegLira has been made by the patient and the treating physician before, which is independent from the decision to participate in this study.
4. Treated with basal insulin plus/minus OADs prior to initiating IDegLira.
5. Available and documented HbA1c measurement below or equal to 12 weeks prior to IDegLira initiation.

Exclusion criteria:

1. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation.
2. Diagnosed with type 1 diabetes mellitus, maturity-onset diabetes of the young, latent autoimmune diabetes in adults, gestational diabetes or any hyperglycaemic state other than T2D.
3. Women known to be pregnant or breastfeeding during the conduct of the study.
4. Patients with basal-bolus insulin prior to IDegLira initiation.
5. Participation in another T2D clinical study that involves any clinical intervention or administration of an investigational drug within 3 months prior to initiating IDegLira.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of male or female adults (above or equal to 18 years at the time of data collection) who are diagnosed with T2D for at least 12 months prior to data collection and were previously treated with basal insulin plus/minus OADs prior to initiating IDegLira. The HbA1c measurement below or equal to 12 weeks prior to IDegLira initiation should be available and documented for each patient to be eligible in the study
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2022-03-22 (Actual); Primary Completion 2022-07-15 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change in local laboratory measured Glycated Haemoglobin A1c (HbA1c) | From baseline (week 0) to end of study (week 26 plus/minus 6 weeks) after IDegLira initiation
  Percentage point

SECONDARY OUTCOMES:
Change in absolute body weight | From baseline (week 0) to end of study (week 26 plus/minus 6 weeks) after IDegLira initiation
  Kilogram (kg)
Comparison between the daily dose of basal insulin and IDegLira | From baseline (week 0) to end of study (week 26 plus/minus 6 weeks) after IDegLira initiation
  Units/day

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (6):
- Colombia (6):
  - Novo Nordisk Investigational Site, Medellín, Antioquia
  - Novo Nordisk Investigational Site, Barranquilla, Atlántico
  - Novo Nordisk Investigational Site, Bogotá, Bogota DC
  - Novo Nordisk Investigational Site, Montería, Departamento de Córdoba
  - Novo Nordisk Investigational Site, Cúcuta, Norte de Santander Department
  - Novo Nordisk Investigational Site, Bucaramanga, Santander Department

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] Ramirez-Rincon A, Henao-Carrillo D, Omeara M, Oliveros J, Assaf J, Ordonez JE, Prasad P, Alzate MA. SPIRIT: Assessing Clinical Parameters Associated with Using IDegLira in Patients with Type 2 Diabetes in a Real-World Setting in Colombia. Diabetes Ther. 2024 Jul;15(7):1535-1545. doi: 10.1007/s13300-024-01593-8. Epub 2024 May 8. PMID 38717577